CLINICAL TRIAL: NCT06893601
Title: The Effect of Parasternal Block on Postoperative Pain in Patients Undergoing Coronary Artery Bypass Graft Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Eray Çağlayan ÇELİk, Principal Investigator, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 97479326-050.04.04
Record Dates: First submitted 2025-03-15; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Postoperative Pain; ICU Hospitalization; Extubation Time
Keywords: Parasternal Block; Postoperative Analgesia; Coronary Artery Bypass Graft Surgery
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Saline group (Placebo Comparator): The saline group received a bilateral parasternal block with 0.9% NaCl solution.
  Interventions: Drug: Parasternal block
- Parasternal block group (Experimental): Parasternal block group, bilateral parasternal block was performed using 0.25% bupivacaine.
  Interventions: Drug: Parasternal block

INTERVENTIONS:
Drug: Parasternal block — A block containing 0.9% NaCl solution was applied to the Saline group just before the sternum was closed by the surgeon, while a bilateral parasternal block using 0.25% bupivacaine was applied to the bupivacaine group. The solutions used for the parasternal block were colorless and indistinguishable to ensure blinding.

SUMMARY:
Objective: This study aims to investigate the effects of intraoperative parasternal block on postoperative analgesia in patients undergoing elective coronary artery bypass graft surgery.

Materials and Methods: This prospective, randomized, double-blind study included 78 patients aged 30-80 years with an ASA (American Society of Anesthesiologists) risk score of III-IV, who were scheduled for elective coronary artery bypass graft surgery. Patients were randomly assigned into two groups: the parasternal block group (n = 39), receiving parasternal block with 2.5% bupivacaine, and the saline group (n = 39), receiving parasternal block with 0.9% NaCl. All patients were administered a standard anesthesia protocol, and routine care and analgesia practices during the postoperative period were not interfered with. Patients in the intensive care unit received intravenous paracetamol every 8 hours for analgesia. If postoperative 24-hour pain scores in the intensive care unit , assessed using the Behavioral Pain Scale while intubated and the Numeric Rating Scale while extubated, exceeded 4, 1 mg/kg tramadol was administered. The timing and doses of the first tramadol administration, as well as extubation times, intensive care unit stay durations, and discharge times, were recorded.

Results: In the postoperative period, Behavioral Pain Scale scores at the 8th hour and Numeric Rating Scale scores at the 4th and 12th hours were significantly lower in the parasternal block group compared to the saline group (p < 0.005). The average extubation time was 8.76 hours in the parasternal block group and 14.76 hours in the saline group (p < 0.001). Among patients with pain scores of 4 or higher, the total tramadol consumption in the parasternal block group was 150 ± 64.72 mg, with the first tramadol administration occurring at 17.26 ± 4.78 hours. In the saline group, total tramadol consumption was 212.5 ± 82.23 mg, and the first administration occurred at 12.35 ± 5.75 hours.

Conclusion: Our study demonstrated that parasternal block, as a component of multimodal analgesia, improved postoperative analgesia levels in coronary artery bypass graft surgery. Therefore, the investigators consider parasternal block to be effective in pain management following median sternotomy.

DETAILED DESCRIPTION:
INTRODUCTION Worldwide, more than 800,000 coronary artery bypass graft surgeries are performed annually. Coronary artery bypass graft surgery is traditionally conducted via median sternotomy, a procedure that can cause damage to both bone and soft tissues. Pain levels are particularly high during the first days following cardiac surgery . Between 30% and 75% of patients report moderate to severe chronic pain after cardiac surgery, and it is known that 4% to 10% develop chronic pain syndrome associated with sternotomy .

Improved pain management reduces surgery-related complications, shortens hospital stays, and enhances patient satisfaction. Traditionally, opioid-based analgesics have been the primary method for postoperative pain control in cardiac surgeries for many years . However, high-dose opioid use is associated with numerous side effects, including sedation, respiratory depression, delayed extubation, urinary retention, itching, nausea, and vomiting . Additionally, intravenous opioid therapy is commonly preferred for postoperative pain management in patients undergoing cardiac surgery.

Thoracic epidural analgesia is a method capable of providing excellent "opioid-free" analgesia following cardiac surgery. Thoracic epidural analgesia has been recognized as an effective alternative due to its ability to reduce respiratory complications, arrhythmias, and mortality rates.

Regional anesthesia, as an essential component of multimodal analgesia approaches, allows cardiac anesthesiologists to minimize opioid consumption. Thoracic epidural and paravertebral blocks are effective methods for continuous pain management; however, their widespread use in cardiac surgery patients is restricted due to the increased risk of epidural hematoma, particularly after cardiac surgery, where coagulopathy, anticoagulation, and antiplatelet drug use are prevalent.

Perioperative analgesic management has become a crucial component of fast-track cardiac anesthesia practices, with the potential to facilitate early tracheal extubation and shorter hospital stays . However, cases where existing pain control methods are insufficient are still observed. In such patients, the use of intravenous opioids during the intraoperative and postoperative periods may lead to undesirable effects such as nausea, vomiting, respiratory depression, and sedation . In this context, parasternal intercostal blocks performed with local anesthetics have been shown to provide adequate analgesia and reduce opioid requirements.

Materials and Methods Ethical Approval This study was approved by the Clinical Research Ethics Committee of Aydın Adnan Menderes University (Ethics Committee Approval Date: January 16, 2020, Decision No: 97479326-050.04.04). The study was conducted in the operating room of Aydın Adnan Menderes University Hospital between February 1, 2020, and February 1, 2021. A total of 80 patients scheduled for elective coronary artery bypass graft surgery and classified as ASA III-IV were included in the study after being appropriately informed and providing verbal and written consent. The study was designed as a prospective, randomized, and double-blind trial.

Randomization

The patients included in the study (n = 80) were divided into two groups according to a randomization sequence prepared in advance by an independent statistician and assigned by the researcher:

1. Parasternal block (PSB) group (n=40)
2. Saline group (n=40) Patients in both groups who were on regular medication for cardiovascular or other systemic diseases continued their usual treatment regimens. The saline group received a block with 0.9% NaCl solution, and paracetamol was administered at 10 mg/kg every eight hours as per the hospital's routine analgesia protocol. In cases of inadequate analgesia, an intravenous infusion of 0.5-1 mg/kg tramadol was added.

In the bupivacaine group, bilateral parasternal block was performed using 0.25% bupivacaine, while in the saline group. The solution used for the parasternal block (local anesthetic or saline) was colorless and indistinguishable. All patients, surgeons, intensive care unit nurses, and outcome assessors were blinded to the treatment allocation Anesthesia Management The patients' age, height, weight, gender, comorbidities, and American Society of Anesthesiologists scores were recorded. Prior to induction in the operating room, a five-lead electrocardiography was used to evaluate heart rhythm, ST-segment changes, and heart rate. Arterial blood pressure was measured via a 20G invasive arterial catheter placed in the radial artery. Peripheral oxygen saturation values were monitored using a pulse oximeter. All these parameters were monitored using a Datex-Ohmeda S/5 anesthesia machine.

All patients received a standard anesthesia protocol. Anesthesia induction for all patients was achieved with 1-1.5 mg/kg propofol, 0.03-0.05 mg/kg midazolam, 3-4 μg/kg fentanyl, 1 mg/kg lidocaine, and 1 mg/kg rocuronium. Following endotracheal intubation, anesthesia maintenance was provided with a 3 L/min flow of a 50/50 O₂/air mixture and 1.5-2% sevoflurane. Using the Seldinger technique under ultrasound guidance, a triple-lumen catheter and a 7F introducer were placed in the right internal jugular vein, and central venous pressure was measured. Body temperature was monitored with an esophageal temperature probe.

Before pericardium incision, patients were administered 300-400 U/kg heparin, and ACT was checked 3 minutes later. The heparin dose was adjusted to maintain an ACT > 480. Intraoperative analgesia was provided with a continuous infusion of fentanyl at a dose of 0.1-0.2 μg/kg/min. Coronary anastomoses were completed under moderate hypothermia (28°C-30°C). After the anastomoses were completed, protamine was administered to antagonize heparin.

At the end of the surgical procedure, just before the closure of the sternotomy, if the patient was in the PSB group according to the randomization, the surgeon administered the prepared 0.25% bupivacaine solution bilaterally into the 2nd to 6th intercostal spaces, 2 cm lateral to the mid-sternal line, beneath the pectoralis major muscle and over the internal intercostal muscle. For the parasternal block, a 20 mL solution was prepared by mixing 10 mL of 0.5% bupivacaine with 10 mL of 0.9% NaCl. From this prepared solution, 2 ml of 0.25% bupivacaine was injected into the parasternal area at each intercostal space, and the procedure was repeated sequentially for 5 levels. The same procedure was performed on the opposite parasternal area. No local anesthetic was applied around the thoracic tube insertion sites. In the saline group, the same procedures were performed using 0.9% NaCl solution.

Postoperative Period After the surgery, the patient was transferred to the intensive care unit while intubated. In the intensive care unit, respiratory support was set to the pressure-controlled synchronized intermittent mandatory ventilation mode. Monitoring of electrocardiogram, peripheral oxygen saturation, invasive arterial pressure, and central venous pressure continued in the intensive care unit. Patients' follow-up in the intensive care unit, extubation times, analgesic use, and transfer from the intensive care unit to the ward were managed according to routine practices. Pain assessment in the intensive care unit was performed and recorded by the intensive care unit nurse responsible for the patient's care. Pain assessment began upon the patient's admission to the intensive care unit and was conducted using the Behavioral Pain Scale at the 1st, 2nd, 4th, and 8th hours while intubated. After extubation, pain was assessed using the Numeric Rating Scale at the 1st, 4th, and 12th hours. During follow-up, if the Behavioral Pain Scale or Numeric Rating Scale scores were 4 or higher and adequate analgesia was not achieved despite the routine administration of 1000 mg paracetamol every eight hours, intravenous tramadol at a dose of 0.5-1 mg/kg was administered.

Paracetamol doses routinely administered every eight hours were not recorded for either group. However, the timing of the first tramadol dose and the total tramadol doses administered were documented from the intensive care unit monitoring charts. Extubation time was defined as the duration between the patient's admission to the intensive care unit and the removal of the endotracheal tube. After extubation, patients' triflo exercise performance, specifically the level of ball elevation (Level 1, 2, 3, or 4), was recorded at the 1st, 4th, and 12th hours. Routine postoperative parameters, including heart rate, cardiac rhythm, SPO₂, blood pressure, and arterial blood gas levels, were recorded. Intensive care unit length of stay and ward length of stay were also documented. Patient satisfaction was assessed in the first postoperative month using the Short Form-36 (SF-36), and the collected data were statistically analyzed.

Statistical Analysis The data were analyzed using the SPSS 19.0 software (IBM, California). An independent samples t-test was used for variables with a normal distribution, while the Mann-Whitney U test was applied for variables not showing a normal distribution. The Pearson Chi-Square test was used for the comparison of categorical data. Statistical significance was defined as p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Study included patients aged 30-80 years
* American Society of Anesthesiologists risk score of III-IV,
* Who were scheduled for elective Coronary Artery Bypass Graft Surgery.

Exclusion Criteria:

* In this study, patients with hypersensitivity to the medications used,
* Patients under 30 years or over 80 years of age,
* Patients with chronic opioid use or severe psychiatric disorders,
* Patients who did not provide informed consent, patients with infection at the injection site,
* Patients with preoperative left ventricular ejection fraction <30%,
* Patients with a history of previous sternotomy,
* Patients with severe renal or liver diseases,
* Patients unable to communicate.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-01-18 (Actual); Primary Completion 2020-10-17 (Actual); Study Completion 2020-10-17 (Actual)

PRIMARY OUTCOMES:
The Effect of Parasternal Block on Postoperative Pain in Patients Undergoing Coronary Artery Bypass Graft Surgery | First 24 Hours in the Intensive Care Unit
  Pain assessment began upon the patient's admission to the ICU and was conducted using the Behavioral Pain Scale at the 1st, 2nd, 4th, and 8th hours while intubated. The lowest score obtained from the scale is 3, and the highest score is 12. An increase in the score indicates an increase in the level of pain.
The Effect of Parasternal Block on Postoperative Pain in Patients Undergoing Coronary Artery Bypass Graft Surgery | First 24 Hours in the Intensive Care Unit
  After extubation, pain was assessed using the Numeric Rating Scale at the 1st, 4th, and 12th hours. Patients report the severity of pain they feel on a scale where 0 indicates no pain and 10 indicates the most severe pain imaginable.

CONTACTS AND LOCATIONS:
Overall Officials: Meryem Nil KAAN, Prof. Dr., Study Director
Locations (1):
- Aydin Adnan Menderes University, Aydin, EFELER, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li Q, Liao Y, Wang X, Zhan M, Xiao L, Chen Y. Efficacy of bilateral catheter superficial parasternal intercostal plane blocks using programmed intermittent bolus for opioid-sparing postoperative analgesia in cardiac surgery with sternotomy: A randomized, double-blind, placebo-controlled trial. J Clin Anesth. 2024 Aug;95:111430. doi: 10.1016/j.jclinane.2024.111430. Epub 2024 Mar 26. PMID 38537393
- [Background] Coriat P, Beaussier M. Fast-tracking after coronary artery bypass graft surgery. Anesth Analg. 2001 May;92(5):1081-3. doi: 10.1097/00000539-200105000-00001. No abstract available. PMID 11323325
- [Background] Schiavoni L, Nenna A, Cardetta F, Pascarella G, Costa F, Chello M, Agro FE, Mattei A. Parasternal Intercostal Nerve Blocks in Patients Undergoing Cardiac Surgery: Evidence Update and Technical Considerations. J Cardiothorac Vasc Anesth. 2022 Nov;36(11):4173-4182. doi: 10.1053/j.jvca.2022.07.025. Epub 2022 Jul 24. PMID 35995636
- [Background] Dogan Baki E, Kavrut Ozturk N, Ayoglu RU, Emmiler M, Karsli B, Uzel H. Effects of Parasternal Block on Acute and Chronic Pain in Patients Undergoing Coronary Artery Surgery. Semin Cardiothorac Vasc Anesth. 2016 Sep;20(3):205-12. doi: 10.1177/1089253215576756. Epub 2015 Apr 21. PMID 25900900
- [Background] Schwann NM, Chaney MA. No pain, much gain? J Thorac Cardiovasc Surg. 2003 Nov;126(5):1261-4. doi: 10.1016/s0022-5223(03)01327-8. No abstract available. PMID 14665993
- [Background] Grant MC, Chappell D, Gan TJ, Manning MW, Miller TE, Brodt JL; PeriOperative Quality Initiative (POQI) and the Enhanced Recovery After Surgery (ERAS) Cardiac Society Workgroup. Pain management and opioid stewardship in adult cardiac surgery: Joint consensus report of the PeriOperative Quality Initiative and the Enhanced Recovery After Surgery Cardiac Society. J Thorac Cardiovasc Surg. 2023 Dec;166(6):1695-1706.e2. doi: 10.1016/j.jtcvs.2023.01.020. Epub 2023 Jan 28. PMID 36868931
- [Background] Hassan S, Stambulic T, King M, Norman P, Payne D, Derry K, et al. Post-Operatıve Paın And Analgesıc Use For Cardıac Surgery Wıth Medıan Sternotomy. Canadian Journal of Cardiology. 2021 Oct 1;37(10):S107-8.
- [Background] Barr AM, Tutungi E, Almeida AA. Parasternal intercostal block with ropivacaine for pain management after cardiac surgery: a double-blind, randomized, controlled trial. J Cardiothorac Vasc Anesth. 2007 Aug;21(4):547-53. doi: 10.1053/j.jvca.2006.09.003. Epub 2006 Dec 22. PMID 17678782
- [Background] Padala SRAN, Badhe AS, Parida S, Jha AK. Comparison of preincisional and postincisional parasternal intercostal block on postoperative pain in cardiac surgery. J Card Surg. 2020 Jul;35(7):1525-1530. doi: 10.1111/jocs.14651. Epub 2020 Jun 24. PMID 32579779
- [Background] Kelava M, Alfirevic A, Bustamante S, Hargrave J, Marciniak D. Regional Anesthesia in Cardiac Surgery: An Overview of Fascial Plane Chest Wall Blocks. Anesth Analg. 2020 Jul;131(1):127-135. doi: 10.1213/ANE.0000000000004682. PMID 32032103
- [Background] Fuchs A, Heinisch PP, Luedi MM, Reid CS. Pain after cardiac surgery: Time to include multimodal pain management concepts in ERAS protocols. J Clin Anesth. 2022 Feb;76:110583. doi: 10.1016/j.jclinane.2021.110583. Epub 2021 Nov 10. No abstract available. PMID 34768206
- [Background] Landoni G, Isella F, Greco M, Zangrillo A, Royse CF. Benefits and risks of epidural analgesia in cardiac surgery. Br J Anaesth. 2015 Jul;115(1):25-32. doi: 10.1093/bja/aev201. PMID 26089444
- [Background] McDonald SB, Jacobsohn E, Kopacz DJ, Desphande S, Helman JD, Salinas F, Hall RA. Parasternal block and local anesthetic infiltration with levobupivacaine after cardiac surgery with desflurane: the effect on postoperative pain, pulmonary function, and tracheal extubation times. Anesth Analg. 2005 Jan;100(1):25-32. doi: 10.1213/01.ANE.0000139652.84897.BD. PMID 15616047
- [Background] Kehlet H, Jensen TS, Woolf CJ. Persistent postsurgical pain: risk factors and prevention. Lancet. 2006 May 13;367(9522):1618-25. doi: 10.1016/S0140-6736(06)68700-X. PMID 16698416
- [Background] Bigeleisen PE, Goehner N. Novel approaches in pain management in cardiac surgery. Curr Opin Anaesthesiol. 2015 Feb;28(1):89-94. doi: 10.1097/ACO.0000000000000147. PMID 25500688
- [Background] Kwanten LE, O'Brien B, Anwar S. Opioid-Based Anesthesia and Analgesia for Adult Cardiac Surgery: History and Narrative Review of the Literature. J Cardiothorac Vasc Anesth. 2019 Mar;33(3):808-816. doi: 10.1053/j.jvca.2018.05.053. Epub 2018 Jun 5. PMID 30064852
- [Background] Huang AP, Sakata RK. [Pain after sternotomy - review]. Rev Bras Anestesiol. 2016 Jul-Aug;66(4):395-401. doi: 10.1016/j.bjan.2014.09.003. Epub 2015 Mar 18. Portuguese. PMID 25796483
- [Background] Reinhart M, Jonsson M, Enthoven P, Westerdahl E. Immediate effects of upper limb exercises with and without deep breathing on lung function after cardiac surgery - a randomized crossover trial. J Cardiothorac Surg. 2024 Aug 28;19(1):503. doi: 10.1186/s13019-024-03007-z. PMID 39198875
- [Background] Nalysnyk L, Fahrbach K, Reynolds MW, Zhao SZ, Ross S. Adverse events in coronary artery bypass graft (CABG) trials: a systematic review and analysis. Heart. 2003 Jul;89(7):767-72. doi: 10.1136/heart.89.7.767. PMID 12807853